CLINICAL TRIAL: NCT06360120
Title: Combining Use of Clopidogrel With Atorvastatin or Rosuvastatin in Patients With Large-vessel Ischemic Stroke, a Randomized Controlled Single-blinded Trial
Brief Title: Combining Use of Clopidogrel With Atorvastatin or Rosuvastatin in Patients With Large-vessel Ischemic Stroke
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed G. zeinhom, MD, principal investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00023098816
Record Dates: First submitted 2024-04-06; First posted 2024-04-11 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke
Keywords: atorvastatin; rosuvastatin; clopidogrel; stroke; Egypt
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Atorvastatin; Tablets; Rosuvastatin Calcium; Clopidogrel

STUDY DESIGN:
Intervention Model Description: The study will be composed of 2 arms atorvastatin arm, which consisted of 300 patients who received 40 mg daily atorvastatin for 3 months, and the rosuvastatin arm consisted of 300 patients who received 20 mg rosuvastatin daily for 3 months, All the patients in the two groups received open-label clopidogrel at a loading dose of 300 mg and then 75 mg daily till the end of the 3 months
Who Masked: Investigator, Outcomes Assessor
Masking Description: Our study was single-blinded to the investigators; an independent statistician generated a computer-generated randomization chart with a block size of four in a one-to-one ratio, and participants were randomly assigned to receive either atorvastatin or rosuvastatin by a specially trained and qualified nurse. None of the investigators included in the study knew the patients' assignments. We prepared Sequentially numbered opaque sealed envelopes and 600 labels for each drug labeled Drug A or B. According to the randomization chart, put them into envelopes numbered 1 to 600. Envelopes were attached to the patient's files. Patients were given enrollment numbers starting from 1, which were mentioned in their files. Files with the same number as the patient enrolment number were opened and the patients were assigned to receive drugs A or B. Drug A included atorvastatin bills, and Drug B included rosuvastatin bills. The statistical analysis was performed by an independent statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- atorvastatin (Active Comparator): The Atorvastatin arm consisted of 300 patients who received 40 mg daily atorvastatin for 3 months, an open-label clopidogrel at a loading dose of 300 mg, and then 75 mg daily till the end of the 3 months
  Interventions: Drug: Atorvastatin 40 Mg Oral Tablet; Drug: Clopidogrel 75 Mg Oral Tablet
- rosuvastatin (Active Comparator): The rosuvastatin arm consisted of 300 patients who received 20 mg daily rosuvastatin for 3 months, an open-label clopidogrel at a loading dose of 300 mg, and then 75 mg daily till the end of the 3 months
  Interventions: Drug: Rosuvastatin 20mg; Drug: Clopidogrel 75 Mg Oral Tablet

INTERVENTIONS:
Drug: Atorvastatin 40 Mg Oral Tablet — The atorvastatin group consisted of 300 patients who received 40 mg daily atorvastatin for 3 months, and open-label clopidogrel at a loading dose of 300 mg and then 75 mg daily till the end of the 3 months.
  Other Names: group A
  Arms: atorvastatin
Drug: Rosuvastatin 20mg — The rosuvastatin group consisted of 300 patients who received 40 mg daily rosuvastatin for 3 months, and open-label clopidogrel at a loading dose of 300 mg and then 75 mg daily till the end of the 3 months.
  Other Names: group B
  Arms: rosuvastatin
Drug: Clopidogrel 75 Mg Oral Tablet — open-label clopidogrel at a loading dose of 300 mg and then 75 mg daily till the end of the 3 months.
  Arms: atorvastatin
Drug: Clopidogrel 75 Mg Oral Tablet — open-label clopidogrel at a loading dose of 300 mg and then 75 mg daily till the end of the 3 months.
  Arms: rosuvastatin

SUMMARY:
Along with the current clinical trial, the impact of adding atorvastatin or rosuvastatin in the first 24 hours on the clinical outcomes of first-ever large-vessel ischemic stroke patients treated with clopidogrel assessed through NIHSS, mRS, and possible adverse effects.

DETAILED DESCRIPTION:
The investigators got written informed consent from all eligible patients or their first order of kin before randomization.

The study will be composed of 2 arms atorvastatin arm, which consisted of 300 patients who received 40 mg daily atorvastatin for 3 months, and the rosuvastatin arm consisted of 300 patients who received 20 mg rosuvastatin daily for 3 months, All the patients in the two groups received open-label clopidogrel at a loading dose of 300 mg and then 75 mg daily till the end of the 3 months.

Study Procedures:

Every patient in our study will undergo:

Clinical workup: History, clinical assessment & NIHSS were recorded on admission, day 7, and the Modified Rankin Scale as a follow-up after one week and 3 months.

Detection of Risk Factors & Profiles:

Echocardiography& TOE: in indicated patients ECG Monitoring: daily ECG monitoring will be performed in indicated patients. - Carotid Duplex: carotid duplex in indicated patients.

4- ESR & Lipid Profile& liver functions: All will be tested routinely for all patients.

Every patient underwent CT brain and MRI brain using stroke protocol: T1W, T2W, FLAIR, DWI, T2 Echo Gradient, CTA, or MRA (if CTA was contraindicated), from the aortic arch through the circle of Willis. Two neuroradiologists blinded to treatment reviewed C.T. and MRI source images. Cerebrovascular vessels were divided into segments: supra-clinoid internal carotid artery, first-division middle cerebral artery (M1), second-division middle cerebral artery (M2), basilar artery (B.A.), intracranial vertebral artery (V.A.). A neuroradiologist determined whether any of these vascular segments were occluded. If there was no vascular occlusion, the patient was documented as having no large vessel occlusion. If one or more vascular segments were occluded and the patient was ineligible for thrombectomy or arterial stenting, the case history and NIHSS score were reviewed; if the vascular occlusion was in the appropriate territory to account for the clinical findings, the case was judged as having a large-vessel occlusion

Primary End Point:

The primary efficacy outcome was the rate of new stroke at 90 days

• Secondary End Point: the secondary efficacy outcomes were to evaluate the rates of patients who achieved a significant reduction in NIHSS (decrease of four points or more) at the seventh day or discharge compared to baseline, the rates of a favorable outcome with (mRS = 0-2) after one week and after 90 days in a face-to-face interview in the outpatient clinic, rates of the composite of recurrent stroke, myocardial infarction, and death due to vascular events after 90 days of follow-up, while the secondary safety outcome was the rate of treatment-related acute liver injury assessed by ALT, AST test at 90 days, statin-induced myopathy assessed by CPK at 90 days and other adverse effects assessed by a follow-up questionnaire.

ELIGIBILITY:
Inclusion Criteria:

- males and females aged 18-75 first-ever large-vessel acute ischemic stroke

Exclusion Criteria:

* the investigators excluded patients with allergies to any of the studied drugs or who suffered from clinical seizures as a part of their stroke, those with major organ failure, malignancies, or myocardial infarction during the past six weeks, and patients who administered regular antiplatelet or anticoagulant in the previous week to avoid clouding our drug safety assessment.
* investigators excluded patients with a minor stroke (National Institutes of Health Stroke Scale (NIHSS) ≤ 3) or severe stroke (NIHSS ≥ 25), patients who had spontaneous resolution of symptoms before imaging, and patients with a history of a CNS disorder (e.g., multiple sclerosis, epilepsy, meningioma).
* investigators excluded Patients were also not eligible if carotid, cerebrovascular, or coronary revascularization was planned, requiring halting study treatment within seven days after randomization.
* investigators excluded Patients who experienced a cardioembolic stroke either prior to or post-treatment were not included in our study. Cardio-embolic strokes were diagnosed when the patient exhibited potential conditions to have a cardiac source of emboli such as mechanical cardiac valves, atrial fibrillation (AF), mitral valve prolapse, aortic valve stenosis or calcification, and patent foramen ovale .
* investigators excluded patients with clinical AF based on the presence of a conventional 12-lead electrocardiography (ECG) recording that exhibited a minimum of 30 seconds of cardiac rhythm, showing the absence of identifiable recurring P waves and irregular RR intervals (when atrioventricular conduction is not impaired).
* investigators excluded patients with a source of gastrointestinal bleeding such as peptic ulcers, patients with recurrent stroke based on appropriate clinical history, examination, and/or MRI brain findings, and those who had a blood glucose level < 50 or > 400 mg/DL or Platelet count < 100,000 or international normalized ratio > 1.4 or Prothrombin time >18.
* investigators excluded patients who were regular users of drugs that affected clopidogrel metabolism, such as proton pump inhibitors, ketoconazole, dihydropyridine calcium channel blockers, and rifampin.
* investigators excluded pregnant or lactating females, patients with venous infarction, and ischemic infarction secondary to hypo-perfusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
the rate of new stroke at 90 days | 90 days
  Rates of new ischemic stroke occur within three months of treatment. The investigators will perform follow-ups of the patient during visits to the outpatient clinic, and brain CT and/ or MRI will be done if there is suspicion of recurrence of ischemic stroke

SECONDARY OUTCOMES:
Value of National Institute of Health Stroke Scale (NIHSS) after one week | 7 days
  NIHSS is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke and aid in planning post-acute care disposition.
  It ranges from 0 to 42; the lower the score, the better the stroke condition. Improvement will be counted only if the NIHSS score decreases by four points or more within one week of stroke onset.
value of Modified Rankin Scale (mRS) at one week | 7 days
  mRS Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability its value ranges from 0 to 6; the lower the score, the better the stroke outcome favorable stroke outcome is considered with mRS value equals two or less.
value of Modified Rankin Scale(mRS) at three months | 3 months
  mRS Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability its value ranges from 0 to 6; the lower the score, the better the stroke outcome favorable stroke outcome is considered with mRS value equals two or less.
rate of composite recurrent stroke, myocardial infarction, and death due to vascular events | 3 months
  rates of new ischemic stroke, TIA, myocardial infarction, or death from vascular events within three months of treatment the investigators will perform follow-ups of the patient during visits to the outpatient clinic and perform needed investigations such as brain imaging, Electrocardiography, arterial and venous duplex ultrasound imaging.
rate of drug adverse effects | 90 days
  Drug adverse effects: all side effects related to the drugs of our study will be reported

CONTACTS AND LOCATIONS:
Overall Officials: mohamed G. Zeinhom, MD, Study Director — neurology department kafr el-sheikh university
Locations (1):
- Kafr Elsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No
All the data that support the findings of this research will be available from the corresponding author M. Zeinhom upon reasonable request.

REFERENCES:
- [Result] Lopez AD, Mathers CD, Ezzati M, Jamison DT, Murray CJ. Global and regional burden of disease and risk factors, 2001: systematic analysis of population health data. Lancet. 2006 May 27;367(9524):1747-57. doi: 10.1016/S0140-6736(06)68770-9. PMID 16731270
- [Result] Zeinhom MG, Aref HM, El-Khawas H, Roushdy TM, Shokri HM, Elbassiouny A. A pilot study of the ticagrelor role in ischemic stroke secondary prevention. Eur Neurol. 2022;85(1):50-55. doi: 10.1159/000518786. Epub 2021 Aug 30. PMID 34515113
- [Result] Paciaroni M, Ince B, Hu B, Jeng JS, Kutluk K, Liu L, Lou M, Parfenov V, Wong KSL, Zamani B, Paek D, Min Han J, Del Aguila M, Girotra S. Benefits and Risks of Clopidogrel vs. Aspirin Monotherapy after Recent Ischemic Stroke: A Systematic Review and Meta-Analysis. Cardiovasc Ther. 2019 Dec 1;2019:1607181. doi: 10.1155/2019/1607181. eCollection 2019. PMID 31867054